CLINICAL TRIAL: NCT06711224
Title: Feasibility Trial of a Guided Internet-delivered Intervention for Adolescents With ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 654423
Record Dates: First submitted 2024-10-01; First posted 2024-12-02 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital intervention (Experimental): The digital intervention includes a mobile app and weekly phone calls with a therapist.
  Interventions: Behavioral: Digital intervention for adolscents with ADHD

INTERVENTIONS:
Behavioral: Digital intervention for adolscents with ADHD — The aim of the digital intervention is to promote coping of ADHD. The intervention has a duration of 6 weeks and will be delivered as a mobile app including weekly phone calls from a therapist. The intervention includes text, interactive exercises, animations, and coping skills. The themes of the intervention includes psychoeducation on ADHD, healthy habits (sleep, exercise, food), social skills, and emotion regulation. The adolescents have the possibility to choose some of the themes they want to work on during the intervention.

SUMMARY:
The main aim of this feasibility trial is to investigate the feasibility and preliminary clinical outcomes of a guided digital intervention for adolescents with ADHD.

Adolescents with ADHD will be enrolled in a 6-week digital intervention including weekly therapist contact. The adolescents and their parents will be asked to complete self-report questionnaires at pre-, during, post- and 3- and 6-months follow-up.

DETAILED DESCRIPTION:
ADHD is one of the most prevalent diagnoses in childhood. Treatment guidelines recommend inclusion of psychological support, however, there are currently few psychological treatment options for adolescents with ADHD.

The current study investigates the feasibility and preliminary effects of therapist-guided digital treatment for adolescents with ADHD using qualitative and quantitative methods. The project uses the person-based approach (PBA) as methodological framework, which is an evidence-based method for developing user-centered and effective behavior change interventions.

The study seeks the examine the intervention within five feasibility domains that includes the following research questions

1. Recruitment 1A. How long does it take to recruit 60 adolescents with ADHD? 1B. Is the target group represented in the sample?
2. Adherence 2A. Does a minimum of 50% complete the intervention? 2B. What characterizes the adolescents who complete the intervention? (predictor) 2C. What characterizes the adolescents who dropout of the intervention? (predictor)
3. Credibility 3A. Will at least 70% of the adolescents recommend the program to a friend with similar challenges?
4. Satisfaction 4A. How satisfied are the adolescents with the intervention? 4B. What are the adolescents' experiences with the intervention? (qualitative feedback)
5. Preliminary clinical outcomes 5A. Will a moderate effect (d = 0.5) on outcomes related to everyday functioning, quality of life and ADHD symptoms be found? 5B. Will more than 40% of the participants experience reliable clinical change (RCI) on the primary clinical outcomes? 5C. Will less than 10% of the participants experience negative clinical effects, defined as a negative RCI?

Youth between the ages of 13 to 16 years and their parents will be invited to participate in this study. The participants will be recruited via child and youth psychiatric outpatient clinics. Eligible participants get access to an online information consent form which is signed digitally using the Norwegian electronic identification system BankID.

Data will be collected using self-report questionnaires administrated online at pre-, during, post- and 3- and 6-months follow-up. The investigators will also conduct semi-structured phone interviews to explore the patients' in-depth experience of the digital treatment. The interviews of approximately 16 adolescents will be conducted 2 to 4 weeks after finishing the treatment. The investigators will strive to have two groups, one with participants that completed the treatment, and one with dropouts.

ELIGIBILITY:
Inclusion criteria:

1. 13-16 years
2. a diagnosis of ADHD
3. parents are willing to participate in answering questionnaires pre, during, post and follow-up
4. stable medication during the study period
5. participant and parents can read, write and speak Norwegian
6. access to mobile phone and internet.

Exclusion criteria:

1. Other primary diagnosis than ADHD (e.g. Autism, intellectual disabilities, severe conduct disorder)
2. clinically significant comorbid psychiatric disorder requiring treatment (e.g. major depression, severe anxiety, suicidal ideation, eating disorder)
3. follows another psychological treatment or intend to start treatment during the intervention period
4. do not follow a regular school plan (e.g. frequently with days away from school/class with different educational content than their peers).

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
The Credibility and Expectancy Scale (CEQ-1) | First week of intervention
  CEQ-1 will be used after participants have completed the first module of the treatment. CEQ measures perceived treatments credibility. The first item "How confident would you be in recommending this treatment to a friend who experiences similar problems?" will be used. The item is rated on a scale from 0 to 10, where higher score indicates better treatment credibility. The question will be administered to the adolescents.
Recruitment rate | From recruitment start and up to 1 year
  The recruitment rate will be assessed by examining number of adolescents recruited per month and total time to recruit 60 adolescents
Satisfaction with intervention | Week 6, at the end of the intervention
  Intervention satisfaction will be measured at post-treatment, using a self-developed questionnaire including 15 items. This questionnaire will be administered to the adolescents.
The strengths and difficulties questionnaire (SDQ) for self-completion | Up to 6-month follow-up
  The strengths and difficulties questionnaire (SDQ) is a questionnaire that consisting of 25 items describing positive and negative attributes of children. Each item is rated on a 3-point scale with response options; not true, somewhat true and certainly true. The questionnaire includes five sub-scales with five items each: 1) emotional symptoms, 2) conduct problems, 3) hyperactivity-inattention problems, 4) peer relationships, and 5) pro-social behavior. The SDQ will be administered to the adolscents. For each of the 5 scales the score can range from 0 to 10 if all items were completed. In addition, a total difficulties score is generated by summing scores from all the scales except the prosocial scale. The resultant score ranges from 0 to 40, where a higher score indicates a higher severity. Lastly, items on overall distress and impairment can be summed to generate an impact score that ranges from 0 to 10, where a higher score indicates higher severity.
KIDSCREEN-10 | Up to 6-month follow-up
  KIDSCREEN-10 is a questionnaire to assess health-related quality of life. The items are rated on 5-point Likert scale that indicates the frequency or intensity of a behavior or emotion. For most items, a higher score reflects higher health-related quality of life. This questionnaire will be administered to the adolescents.
Module completion | From intervention start and up to 6 weeks.
  Number of modules completed will be used to assess adherence to the intervention.
Time spent in app | From intervention start and up to 6 weeks.
  The time spent in the app will be used to assess adherence
Logins to app | From intervention start and up to 6 weeks.
  Number of logins to the app will be used to assess adherence to the intervention
The strengths and difficulties questionnaire (SDQ) for parents | Up to 6-month follow-up
  The strengths and difficulties questionnaire (SDQ) is a questionnaire that consisting of 25 items describing positive and negative attributes of children. Each item is rated on a 3-point scale with response options; not true, somewhat true and certainly true. The questionnaire includes five sub-scales with five items each: 1) emotional symptoms, 2) conduct problems, 3) hyperactivity-inattention problems, 4) peer relationships, and 5) pro-social behavior. For each of the 5 scales the score can range from 0 to 10 if all items were completed. In addition, a total difficulties score is generated by summing scores from all the scales except the prosocial scale. The resultant score ranges from 0 to 40, where a higher score indicates a higher severity. Lastly, items on overall distress and impairment can be summed to generate an impact score that ranges from 0 to 10, where a higher score indicates higher severity.

SECONDARY OUTCOMES:
UCLA loneliness scale | Up to 6 months follow-up
  UCLA loneliness scale measures subjective feelings of loneliness and social isolation. The questionnaire is a 20 item scale where participants rate either O ("I often feel this way"), S ("I sometimes feel this way"), R ("I rarely feel this way"), N ("I never feel this way"). The total score ranges from 20 to 80. Higher scores indicate higher loneliness. The scale will be administered to the adolescents.
Knowledge on ADHD | Week 6, at the end of the intervention
  Knowledge on ADHD: The adolescents will be asked: "do you experience increased knowledge about ADHD after participating in this program?" as a part of the post-treatment assessment. The response options will include: "not at all", "to a small extent" "to some extent", to a good extent" and "to a large extent".
Mood | From intervention start and up to week 6.
  As a part of the intervention, the adolescents will be asked to rate their mood daily in the mobile app using cartoons with response options ranging from "awful", "not so good", "okay", "pretty good" and "amazing".
Sleep, eating and exercise habits | Up to 6 months follow-up
  As a part of the 3 module, the adolescents will be asked to either rate of their sleep, eating or exercise habits on daily basis. They will be asked how satisfied they with their eating / sleeping / exercise habits on a scale from 1 (Very dissatisfied) to 5 (Very satisfied) and how much their eating / sleeping / exercise habits is affecting their daily functioning on a scale from 1 (Not at all) to 5 (Very much). The adolescents choose themselves what area (eating, sleeping or exercise habits) they want to focus on. In addition, the adolescents will be asked these questions at pre, post and follow-up.
SNAP IV 18 | Up to 6 months follow-up
  The Norwegian version of the SNAP-IV 18 consists of the 18 symptoms for ADHD as described by the DSM-IV. The scale includes on inattention subscale and one hyperactivity subscale. Responses are rated on a 4-point scale with response options: not at all/just a little bit/quite a bit/very much. Subscale scores on the SNAP-IV are calculated by summing the scores on the items in the subset and dividing by the number of items in the subset. The score for any subset is expressed as the Average Rating-Per-Item. The questionnaire will be administered to parents at pre, post, and 3 and 6 months after the treatment.
Difficulties in Emotion Regulation Scale (DERS) | Up to 6-month follow-up
  Difficulties in Emotion Regulation Scale (DERS) measures emotion regulation problems. The study will apply the short version containing 16 items with the following sub-scales: nonacceptance of emotional responses; difficulty engaging in goal-directed behaviour; impulse control difficulties; lack of emotional awareness; limited access to emotion regulation strategies; lack of emotional clarity. The total score ranges from 16-80 with higher scores indicating more difficulties with emotion regulation. This questionnaire will be administered to the adolescents.

OTHER OUTCOMES:
The readiness to change questionnaire (RTCQ-6) | Baseline
  The readiness to change questionnaire (RTCQ-6) is adapted to the study population and digital treatment inspired by the Short Motivation Feedback List (SMFL-8). The questionnaire will be administered to the adolescents.
Self-efficacy | Baseline
  A Self-efficacy (SE) scale consisting of 15 items will be administered to the adolescents pre intervention to investigate their belief in their own ability to use the intervention.
ADHD among relatives | Baseline
  ADHD among relatives will be assessed by asking: How many in the adolescents' close family (siblings, parents, grandparents, uncles, aunts or cousins) have an ADHD diagnosis? The question will be administered to the parents.

CONTACTS AND LOCATIONS:
Overall Officials: Tine Nordgreen, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No